CLINICAL TRIAL: NCT01090882
Title: Efficacy of Intraperitoneal Local Anaesthetic Techniques During Laparoscopic Cholecystectomy: A Double Blind Randomized Controlled Trial
Brief Title: Intraperitoneal Techniques of Local Anaesthesia During Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHCW 1
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Gall Stones
Keywords: Local anaesthetic; Laparoscopic cholecystectomy; Pain scores; Bupivocaine; Day case surgery
MeSH Terms: conditions — Gallstones | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Sham Comparator): Sham wash, sham injection
  Interventions: Drug: 0.9% normal saline solution
- Subperitoneal injection (Experimental): Local anaesthetic injection to diaphragm with sham wash over liver and gall bladder
  Interventions: Drug: Bupivocaine
- Topical LA (Active Comparator): Local anaesthetic washed over gall bladder and liver. Sham injection of diaphragm
  Interventions: Drug: Bupivocaine

INTERVENTIONS:
Drug: Bupivocaine — 20ml 0.25% at beginning of operation
  Other Names: marcaine
  Arms: Subperitoneal injection; Topical LA
Drug: 0.9% normal saline solution — 20ml 0.9% NaCl
  Other Names: marcaine
  Arms: Control

SUMMARY:
Pain following laparoscopic cholecystectomy (LC) results in morbidity and is a barrier to same day discharge. In several trials local anaesthetic (LA) washed over the liver and gall bladder decreases pain. In many patients pain has a strong component attributable to diaphragmatic origin. A wash of LA over the liver and gall bladder is unlikely to provide high levels of analgesia to pain fibres from the diaphragm. The investigators hypothesise that LA injected to the right hemidiaphragm during LC would be more effective than wash.

Methods Double blind randomised controlled trial of 128 consecutive subjects undergoing elective LC. Control -sham injection of diaphragm and sham wash over liver/GB with saline; Test treatment 'subperitoneal LA' - bupivocaine injection/sham wash; Internal control 'topical LA' - sham injection/bupivocaine wash. Primary outcome: pain scores in theatre recovery and the ward. Secondary outcomes: analgesic use, physiological observations, time to eating and mobilising, day case surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy
* 18 years old or over

Exclusion Criteria:

* Emergency surgery
* Under 18 year olds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
VAS pain score | 1, 4, 8 hours after operation and at discharge

SECONDARY OUTCOMES:
Time to ambulation | following the procedure
  The first time the patient gets out of bed and walks following the procedure
Same day discharge | 24 hours
VRS pain scores | Every 10 minutes in theatre recovery
  Immediately following the operation

CONTACTS AND LOCATIONS:
Overall Officials: Keith J Roberts, MRCS, Principal Investigator — University Hospital Coventry and Warwickshire NHS Trust
Locations (1):
- UHCW NHS Trust, Coventry, Warwickshire, United Kingdom

REFERENCES:
- [Derived] Roberts KJ, Gilmour J, Pande R, Nightingale P, Tan LC, Khan S. Efficacy of intraperitoneal local anaesthetic techniques during laparoscopic cholecystectomy. Surg Endosc. 2011 Nov;25(11):3698-705. doi: 10.1007/s00464-011-1757-3. Epub 2011 Jun 3. PMID 21638181